CLINICAL TRIAL: NCT00601419
Title: Drug Use Investigation of GENOTROPIN for GHD-ADULTS.
Brief Title: Drug Use Investigation of Somatropin for GHD-ADULTS.
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6281286
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Results first posted 2014-02-06 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2013-12

CONDITIONS: Dwarfism, Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Somatropin: Patients administered Somatropin.
  Interventions: Drug: Somatropin

INTERVENTIONS:
Drug: Somatropin — Genotropin® 12mg for Injection, Genotropin® MiniQuick for s.c. injection 0.6mg, Genotropin® MiniQuick for s.c. injection 1.0mg, Genotropin® MiniQuick for s.c. injection 1.4mg, Genotropin® 5.3mg.
  Dosage, Frequency: According to Japanese LPD, "The initial dosage is 0.021mg/kg/week as somatropin (genetical recombination) in 6-7 divided doses by s.c. route. The dosage is titrated by 0.084mg/kg/week at a maximum according to the patient's clinical symptoms, and administered in 6-7 divided doses in a week by s.c. route. The dosage may be adjusted according to patient's clinical symptoms and laboratory test results such as serum Insulin-like Growth Factor-I (IGF-I) concentrations. However, the maximum daily dosage shouldn't be higher than 1mg/day".
  Duration: According to the protocol of A6281286, the duration of the investigation for findings regarding safety and efficacy of a patient is from the first drug administration to the 6 month after the first administration.

SUMMARY:
Post marketing drug use investigation of Genotropin for GHD-ADULTS.

DETAILED DESCRIPTION:
All the patients whom an investigator prescribes the first Somatropin should be registered consecutively until the number of subjects reaches target number.

ELIGIBILITY:
Inclusion Criteria:

The patients who were administered Somatropin to treat "Adult growth hormone deficiency (limited to severe type)".

Exclusion Criteria:

Patients not administered Somatropin.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients whom an investigator involving A6281286 prescribes the Somatropin.
Sampling Method: Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2007-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- [Derived] Morrhaye G, Kermani H, Legros JJ, Baron F, Beguin Y, Moutschen M, Cheynier R, Martens HJ, Geenen V. Impact of growth hormone (GH) deficiency and GH replacement upon thymus function in adult patients. PLoS One. 2009 May 22;4(5):e5668. doi: 10.1371/journal.pone.0005668. PMID 19479077
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6281286&StudyName=Drug%20Use%20Investigation%20of%20Somatropin%20for%20GHD-ADULTS.

RESULTS

PARTICIPANT FLOW:
Groups:
- Somatropin: Participants taking somatropin for adult growth hormone deficiency according to Japanese package insert.
Period: Overall Study
Arm/Group | Somatropin
Started | 230
Completed | 226
Not Completed | 4
Not completed — Lost to Follow-up | 3
Not completed — Missed Visits | 1

BASELINE CHARACTERISTICS:
Arm/Group | Somatropin
Number analyzed (Participants) | 226
Age, Customized [Number; unit: participants]
  <65 years | 196
  >=65 years | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120
  Male | 106

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Related Adverse Events.
Description: Adverse events mean all unfavorable events that occur in participants after administration of somatropin, irrespective of causal relationship to somatropin (including clinically problematic abnormal changes in laboratory test values). Treatment related adverse events were evaluated in company with the causal relationship to somatropin.
Time Frame: 6 month
Population: The safety analysis population consists of the participants who satisfy the case conditions and in whom administration of this drug was confirmed.
Measure: Number; unit: participants
Arm/Group | Somatropin
Number analyzed (Participants) | 226
participants | 29

2. Primary Outcome: Number of Unlisted Treatment Related Adverse Events According to Japanese Package Insert.
Description: Adverse events mean all unfavorable events that occur in participants after administration of somatropin, irrespective of causal relationship to somatropin (including clinically problematic abnormal changes in laboratory test values). Treatment related adverse events were evaluated in company with the causal relationship to somatropin. Unlisted treatment related adverse events were confirmed with listed adverse drug reaction according to Japanese package insert.
Time Frame: 6 month
Population: as for outcome 1
Measure: Number; unit: events
Arm/Group | Somatropin
Number analyzed (Participants) | 226
events | 8

3. Primary Outcome: Number of Participants With Treatment Related Adverse Events of Somatropin: <65 Years of Age vs. >=65 Years of Age.
Description: To determine whether age is a significant risk factor in the frequency of treatment related adverse events.
Time Frame: 6 month
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- <65 Years: Participants younger than 65 years of age when taking somatropin for adult growth hormone deficiency according to Japanese package insert.
- >=65 Years: Participants older than or equal to 65 years of age when taking somatropin for adult growth hormone deficiency according to Japanese package insert.
Arm/Group | <65 Years | >=65 Years
Number analyzed (Participants) | 196 | 30
participants | 24 | 5
Statistical Analysis 1: Comparison: <65 Years vs >=65 Years; The risk factor tested was "Age". The null hypothesis is that there is no difference between "<65 years and >=65 years" in the frequency of treatment related adverse events; Test type: Superiority or Other; p = 0.556, Fisher Exact

4. Primary Outcome: Number of Participants With Treatment Related Adverse Events of Somatropin by Gender.
Description: To determine whether gender is a significant risk factor in the frequency of treatment related adverse events.
Time Frame: 6 month
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Male: Male participants taking somatropin for adult growth hormone deficiency according to Japanese package insert.
- Female: Female participants taking somatropin for adult growth hormone deficiency according to Japanese package insert.
Arm/Group | Male | Female
Number analyzed (Participants) | 106 | 120
participants | 13 | 16
Statistical Analysis 1: Comparison: Male vs Female; The risk factor tested was "Gender". The null hypothesis is that there is no difference between "Male and Female" in the frequency of treatment related adverse events; Test type: Superiority or Other; p = 0.845, Fisher Exact

5. Primary Outcome: Number of Participants With Treatment Related Adverse Events of Somatropin: With Thyroid Stimulating Hormone (TSH) Deficiency vs. Without TSH Deficiency.
Description: To determine whether TSH deficiency is a significant risk factor in the frequency of treatment related adverse events.
Time Frame: 6 month
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Participants With TSH Deficiency: Participants with TSH deficiency taking somatropin for adult growth hormone deficiency according to Japanese package insert.
- Participants Without TSH Deficiency: Participants without TSH deficiency taking somatropin for adult growth hormone deficiency according to Japanese package insert.
Arm/Group | Participants With TSH Deficiency | Participants Without TSH Deficiency
Number analyzed (Participants) | 169 | 56
participants | 17 | 12
Statistical Analysis 1: Comparison: Participants With TSH Deficiency vs Participants Without TSH Deficiency; The null hypothesis is that there is no difference between "With TSH deficiency and Without TSH deficiency" in the frequency of treatment related adverse events; Test type: Superiority or Other; p = 0.038, Fisher Exact

6. Primary Outcome: Number of Participants With Treatment Related Adverse Events of Somatropin: With Past History of Any Disease vs. Without Past History of Any Disease.
Description: To determine whether past history of any disease is a significant risk factor in the frequency of treatment related adverse events.
Time Frame: 6 month
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Participants With Past History of Any Disease: Participants with past history of any disease taking somatropin for adult growth hormone deficiency according to Japanese package insert.
- Participants Without Past History of Any Disease: Participants without past history of any disease taking somatropin for adult growth hormone deficiency according to Japanese package insert.
Arm/Group | Participants With Past History of Any Disease | Participants Without Past History of Any Disease
Number analyzed (Participants) | 143 | 83
participants | 17 | 12
Statistical Analysis 1: Comparison: Participants With Past History of Any Disease vs Participants Without Past History of Any Disease; The risk factor tested was "Past history". The null hypothesis is that there is no difference between "With past history and Without past history" in the frequency of treatment related adverse events; Test type: Superiority or Other; p = 0.013, Fisher Exact

7. Primary Outcome: Number of Participants With Treatment Related Adverse Events of Somatropin by Initial Dose of Somatropin.
Description: To determine whether initial dose of somatropin is a significant risk factor in the frequency of treatment related adverse events.
Time Frame: 6 month
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- <0.021 mg/kg/Week: Participants taking an initial dose of less than 0.021 mg/kg/week of somatropin for adult growth hormone deficiency according to Japanese package insert.
- >=0.021 mg/kg/Week and <0.042 mg/kg/Week: Participants taking an initial dose of 0.021 mg/kg/week or more and less than 0.042 mg/kg/week of somatropin for adult growth hormone deficiency according to Japanese package insert.
- >=0.042 mg/kg/Week and <=0.084 mg/kg/Week: Participants taking an initial dose of 0.042 mg/kg/week or more and 0.084 mg/kg/week or less of somatropin for adult growth hormone deficiency according to Japanese package insert.
- >0.084 mg/kg/Week: Participants taking an initial dose of more than 0.084 mg/kg/week of somatropin for adult growth hormone deficiency according to Japanese package insert.
Arm/Group | <0.021 mg/kg/Week | >=0.021 mg/kg/Week and <0.042 mg/kg/Week | >=0.042 mg/kg/Week and <=0.084 mg/kg/Week | >0.084 mg/kg/Week
Number analyzed (Participants) | 133 | 80 | 5 | 5
participants | 23 | 4 | 0 | 1
Statistical Analysis 1: Comparison: <0.021 mg/kg/Week vs >=0.021 mg/kg/Week and <0.042 mg/kg/Week vs >=0.042 mg/kg/Week and <=0.084 mg/kg/Week vs >0.084 mg/kg/Week; The risk factor tested was "Initial Dose". The null hypothesis is that there is no association between "Initial Dose and the frequency of treatment related adverse events"; Test type: Superiority or Other; p = 0.037, Fisher Exact
Statistical Analysis 2: Comparison: <0.021 mg/kg/Week vs >=0.021 mg/kg/Week and <0.042 mg/kg/Week vs >=0.042 mg/kg/Week and <=0.084 mg/kg/Week vs >0.084 mg/kg/Week; The risk factor tested was "Initial Dose". The null hypothesis is that there is no linear trend in the frequency of treatment related adverse events across increasing levels of initial dose; Test type: Superiority or Other; p = 0.063, Cochran-Armitage Exact

8. Primary Outcome: Proportion of Participants Achieving Clinical Efficacy.
Description: Number of participants achieving clinical efficacy / Number of evaluable participants. Clinical efficacy was assessed comprehensively by physicians in three categories, 'effective', 'not effective', and 'not evaluable', based on the time profile of variables.
Time Frame: 6 month
Population: The efficacy analysis population basically consists of the evaluable participants in whom clinical responses were assessed comprehensively based on the time profile of variables including IGF-I, blood pressures, pulse rate, lipid metabolism, body composition, QOL, and degree of participant's satisfaction.
Measure: Number; unit: participants
Arm/Group | Somatropin
Number analyzed (Participants) | 199
participants
  Effective | 185
  Not effective | 14
  Not evaluable | 0

9. Primary Outcome: Proportion of Participants Achieving Clinical Efficacy: <65 Years of Age vs. >=65 Years of Age.
Description: as for outcome 8
Time Frame: 6 month
Population: as for outcome 8
Measure: Number; unit: participants
Groups:
- <65 Years: Participants younger than 65 years of age while taking somatropin for adult growth hormone deficiency according to Japanese package insert.
- >=65 Years: Participants older than or equal to 65 years of age while taking somatropin for adult growth hormone deficiency according to Japanese package insert.
Arm/Group | <65 Years | >=65 Years
Number analyzed (Participants) | 174 | 25
participants | 165 | 20
Statistical Analysis 1: Comparison: <65 Years vs >=65 Years; The risk factor tested was "Age". The null hypothesis is that there is no difference between "<65 years of age and >=65 years of age" in the efficacy of somatropin"; Test type: Superiority or Other; p = 0.019, Fisher Exact

10. Primary Outcome: Proportion of Participants Achieving Clinical Efficacy by Gender.
Description: as for outcome 8
Time Frame: 6 month
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Male | Female
Number analyzed (Participants) | 92 | 107
participants | 86 | 99
Statistical Analysis 1: Comparison: Male vs Female; The risk factor tested was "Gender". The null hypothesis is that there is no difference between "male and female" in the efficacy of somatropin"; Test type: Superiority or Other; p = 1.000, Fisher Exact

11. Primary Outcome: Proportion of Participants Achieving Clinical Efficacy: With ACTH Deficiency vs. Without ACTH Deficiency.
Description: as for outcome 8
Time Frame: 6 month
Population: as for outcome 8
Measure: Number; unit: participants
Groups:
- Participants With ACTH Deficiency: Participants with ACTH deficiency taking somatropin for adult growth hormone deficiency according to Japanese package insert.
- Participants Without ACTH Deficiency: Participants without ACTH deficiency taking somatropin for adult growth hormone deficiency according to Japanese package insert.
Arm/Group | Participants With ACTH Deficiency | Participants Without ACTH Deficiency
Number analyzed (Participants) | 128 | 67
participants | 116 | 66
Statistical Analysis 1: Comparison: Participants With ACTH Deficiency vs Participants Without ACTH Deficiency; The risk factor tested was "ACTH deficiency". The null hypothesis is that there is no difference between "With ACTH deficiency and Without ACTH deficiency" in the efficacy of somatropin"; Test type: Superiority or Other; p = 0.037, Fisher Exact

ADVERSE EVENTS:
Description: The frequency of treatment related adverse events.
Arm/Group | Somatropin
Serious Adverse Events (participants affected / at risk) | 10/226
Other Adverse Events (participants affected / at risk) | 19/226
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Somatropin (N=226)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Craniopharyngioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Germ cell cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Intraocular pressure increased (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Somatropin (N=226)
Pneumonia (Infections and infestations) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Feeling abnormal (General disorders) | 1 (1)
Injection site haemorrhage (General disorders) | 2 (2)
Oedema (General disorders) | 2 (2)
Oedema peripheral (General disorders) | 1 (1)
Insulin-like growth factor increased (Investigations) | 1 (1)
Blood cholesterol increased (Investigations) | 1 (1)
Blood triglycerides increased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.